CLINICAL TRIAL: NCT00743119
Title: Comparison of the Analgesic Effects of Dronabinol and Smoked Marijuana in Daily Marijuana Smokers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Research Foundation for Mental Hygiene, Inc. (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 5603; 5P50DA009236 (NIH)
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Results first posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Pain Threshold; Mood
Keywords: oral thc; cannabis; pain; analgesic effects; dronabinol
MeSH Terms: conditions — Marijuana Abuse; Pain | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Placebo-controlled, double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo + inactive marijuana (0% THC) (Placebo Comparator): Participants received placebo capsules and smoked inactive marijuana (0% THC) on 1 of 5 outpatient sessions in randomized order.
  Interventions: Drug: Placebo capsules; Drug: Inactive marijuana (0% THC)
- Dronabinol 10 mg + Marijuana (0% THC) (Experimental): Participants received low dose Dronabinol + inactive marijuana (0% THC) on 1 of 5 outpatient sessions in randomized order.
  Interventions: Drug: Inactive marijuana (0% THC); Drug: Low dose Dronabinol
- Dronabinol 20 mg + Marijuana (0% THC) (Experimental): Participants received High dose Dronabinol + inactive marijuana (0% THC) on 1 of 5 outpatient sessions in randomized order.
  Interventions: Drug: Inactive marijuana (0% THC); Drug: High dose Dronabinol
- Placebo + Marijuana (1.98% THC) (Experimental): Participants received placebo + low THC marijuana (1.98% THC) on 1 of 5 outpatient sessions in randomized order.
  Interventions: Drug: Placebo capsules; Drug: Low THC marijuana
- Placebo + Marijuana (3.56% THC) (Experimental): Participants received placebo + smoked high THC marijuana (3.56 % THC) on 1 of 5 outpatient sessions in randomized order.
  Interventions: Drug: Placebo capsules; Drug: High THC marijuana

INTERVENTIONS:
Drug: Placebo capsules — Placebo capsules
  Arms: Placebo + Marijuana (1.98% THC); Placebo + Marijuana (3.56% THC); Placebo + inactive marijuana (0% THC)
Drug: Inactive marijuana (0% THC) — Inactive marijuana cigarettes (0% THC) provided by NIDA
  Arms: Dronabinol 10 mg + Marijuana (0% THC); Dronabinol 20 mg + Marijuana (0% THC); Placebo + inactive marijuana (0% THC)
Drug: Low dose Dronabinol — Dronabinol 10mg
  Arms: Dronabinol 10 mg + Marijuana (0% THC)
Drug: High dose Dronabinol — Dronabinol 20mg
  Arms: Dronabinol 20 mg + Marijuana (0% THC)
Drug: Low THC marijuana — marijuana cigarettes (1.98% THC) provided by NIDA
  Arms: Placebo + Marijuana (1.98% THC)
Drug: High THC marijuana — Marijuana cigarettes (3.56% THC) provided by NIDA
  Arms: Placebo + Marijuana (3.56% THC)

SUMMARY:
The following study is designed to determine the analgesic efficacy of smoked marijuana (0, 1.98, and 3.56% THC) and oral THC (0, 10, and 20 mg) in the Cold-Pressor Test (CPT), a laboratory model of pain which has predictive validity for clinical use of analgesics. Oral THC (dronabinol) is known to have a slower onset and longer duration of action compared with smoked marijuana. Therefore, the analgesic effects of oral THC is expected to peak later and last longer than effects produced by smoked marijuana.

DETAILED DESCRIPTION:
Laboratory animal studies have demonstrated the analgesic effects of drugs which act on the cannabinoid system, however, these effects have et to be clearly elucidated in humans. To better understand the potential clinical application of cannabinoids for pain management, the following study is designed to determine the analgesic efficacy of smoked marijuana (3.56% THC) and oral THC (20 mg) in the Cold-Pressor Test (CPT), a laboratory model of pain which has predictive validity for clinical use of analgesics. Non-treatment seeking marijuana smokers will be recruited for a five-session study during which the analgesic, subjective, and physiologic effects of cannabinoids will be evaluated. Determining the efficacy of cannabinoids in an experimental model of pain will provide important endpoints (i.e., dose, route of administration, time course) or this effect to further investigate the potential role for clinical use of smoked marijuana and/or oral THC as analgesics.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 21-45
* Current marijuana use
* Able to perform study procedures
* Women practicing an effective form of birth control

Exclusion Criteria:

* Female subjects who are currently pregnant or breastfeeding
* Current,repeated illicit drug use other than marijuana
* Presence of significant medical illness
* History of heart disease
* Request for drug treatment
* Current parole or probation
* Recent history of significant violent behavior

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2008-06; Primary Completion 2009-10 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Haney, Ph.D, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cooper ZD, Comer SD, Haney M. Comparison of the analgesic effects of dronabinol and smoked marijuana in daily marijuana smokers. Neuropsychopharmacology. 2013 Sep;38(10):1984-92. doi: 10.1038/npp.2013.97. Epub 2013 Apr 22. PMID 23609132

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirty-four participants were enrolled, and 30 completed. A total of 30 participants completed all 5 treatment combinations in randomized order.
Groups:
- Placebo/Dronabinol + Marijuana: During each session, one capsule containing placebo or dronabinol (10 mg or 20 mg) was administered to the participant 45 min before marijuana was smoked (0, 1.98, or 3.56% THC marijuana). Only one active dose of marijuana or dronabinol was administered within a session. A within-subject design was used in which all participants received all strengths of dronabinol and marijuana. The order was randomized.
Period: Overall Study
Arm/Group | Placebo/Dronabinol + Marijuana
Started | 34
Completed | 30
Not Completed | 4
Not completed — unreliable | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall Number of Baseline Participants: 34 participants were enrolled, but only 30 participants completed. Out of the additional 4 volunteers, 1 discontinued for personal reasons and three were unreliable.
Arm/Group | Overall Number of Baseline Participants
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Pain Tolerance
Description: Change in pain tolerance from baseline (in seconds) as a function of drug condition. The cold pressor test was administered during each session to examine changes in pain threshold (how many seconds it takes for a participant to begin feeling pain after cold water immersion).
Time Frame: Within each session lasting approximately 5 minutes, for a total of five sessions
Population: All participants who completed the study (N=30) were included in the final analysis.
Measure: Mean (Standard Error); unit: seconds
Groups:
- High Dose Dronabinol + Inactive Marijuana: Dronabinol 20 mg + inactive marijuana (0%THC)
- Low Dose Dronabinol + Inactive Marijuana: 10mg Dronabinol + inactive Marijuana (0% THC)
- Placebo + Low THC Marijuana: Placebo + Marijuana (1.98% THC)
- Placebo + High THC Marijuana: Placebo + high dose Marijuana (3.56% THC)
- Placebo + Inactive Marijuana 0% THC: Placebo + inactive marijuana (0% THC)
Arm/Group | High Dose Dronabinol + Inactive Marijuana | Low Dose Dronabinol + Inactive Marijuana | Placebo + Low THC Marijuana | Placebo + High THC Marijuana | Placebo + Inactive Marijuana 0% THC
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 30
seconds | 6.1 (4.4) | 2.8 (2.9) | 4.9 (3.4) | 1.5 (1.4) | 1.5 (1.4)

ADVERSE EVENTS:
Time Frame: Adverse events were documented pre- and post-treatment and 1 week after completion of the entire study.
Description: Research staff routinely asked participants to report any adverse events occurring during study sessions and during outpatient washout periods.
Groups:
- Placebo + Marijuana (0% THC): Adverse events recorded during Placebo (PBO) + Marijuana (0% THC) treatment
- Dronabinol 10 mg + Marijuana (0% THC): Adverse events recorded during Dronabinol 10 mg + Marijuana (0% THC) treatment
- Dronabinol 20mg + Marijuana (0% THC): Adverse events recorded during Dronabinol 20mg + Marijuana (0% THC) treatment
- Placebo + Marijuana (1.98% THC): Adverse events recorded during placebo + Marijuana (1.98% THC) treatment
- Placebo + Marijuana (3.56% THC): Adverse events recorded during Placebo + Marijuana (3.56% THC) treatment
Arm/Group | Placebo + Marijuana (0% THC) | Dronabinol 10 mg + Marijuana (0% THC) | Dronabinol 20mg + Marijuana (0% THC) | Placebo + Marijuana (1.98% THC) | Placebo + Marijuana (3.56% THC)
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34 | 0/34 | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/34 | 0/34 | 0/34 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No